CLINICAL TRIAL: NCT03062618
Title: Randomized, Double Blind, Placebo Controlled, Incomplete Crossover Single Oral Dose Escalation of PRCL-02 in Normal Healthy Volunteers (Part A) and Multiple Oral Dose Escalation in Normal Healthy Volunteers (Part B) and in Chronic Plaque Psoriasis Patients (Part C)
Brief Title: A Study of PRCL-02 in Healthy Volunteers and Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PRCL Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRCL-SMAD
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part A: Single Dose (Experimental): Two escalating sequences of single oral doses of PRCL-02, in 3 periods, starting at 4 milligrams (mg)
  Interventions: Drug: PRCL-02
- Part A: Single Dose (Placebo) (Placebo Comparator): Two escalating sequences of matching placebo oral tablets, in 3 periods
  Interventions: Drug: Placebo Oral Tablet
- Part B: Multiple Dose (Experimental): Multiple oral doses of PRCL-02 for 28 days, at up to 3 dose levels
  Interventions: Drug: PRCL-02
- Part B: Multiple Dose (Placebo) (Placebo Comparator): Multiple oral doses of placebo for 28 days, at matching dose levels
  Interventions: Drug: Placebo Oral Tablet
- Part C: Multiple Dose (Experimental): Multiple oral doses of PRCL-02 for 28 days, at up to 3 dose levels
  Interventions: Drug: PRCL-02
- Part C: Multiple Dose (Placebo) (Placebo Comparator): Multiple oral doses of placebo for 28 days, at matching dose levels
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: PRCL-02 — Oral tablet(s) administered with water
  Arms: Part A: Single Dose; Part B: Multiple Dose; Part C: Multiple Dose
Drug: Placebo Oral Tablet — Administered with water
  Arms: Part A: Single Dose (Placebo); Part B: Multiple Dose (Placebo); Part C: Multiple Dose (Placebo)

SUMMARY:
This study consists of three parts: single oral dose escalation in healthy volunteers (Part A), and multiple oral dose escalations in healthy volunteers (Part B) and in participants with chronic plaque psoriasis (Part C)

ELIGIBILITY:
Inclusion Criteria:

Parts A and B

* Be 18 to 55 years old
* Be healthy with absence of clinically significant illness
* Male participants must agree to use medically accepted methods of contraception with all sexual partners during the study, and for 90 days after
* Female participants must be postmenopausal or surgically sterile
* Have venous access sufficient for blood sampling
* Be a non-smoker

Part C

* Be 18 to 75 years old
* Have chronic plaque psoriasis based on a confirmed diagnosis of plaques for at least 6 months
* Have at least 2 evaluable plaques located in at least 2 body regions

Exclusion Criteria:

Parts A and B

* Significant abnormalities in vital signs, laboratory tests, electrocardiogram, or history of heart disease, some allergies, or infections
* Hepatic or renal impairment
* Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV)
* Female participants who are pregnant or breast feeding
* Recent or ongoing infection
* History of alcohol or drug abuse
* Current or recent enrollment in a clinical trial judged not compatible with this study

Part C

* Have highly active psoriatic arthritis
* Have pustular, erythrodermic and/or guttate forms of psoriasis
* Have had a clinically-significant flare of psoriasis during the last 12 weeks
* Currently or recently taking certain prescribed therapies for psoriasis
* Use of selected topical treatments within 4 weeks prior to starting the study (use of some emollients without urea is allowed, except on one lesion for biopsy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Events (Part A) | Baseline up to approximately 45 days
  Number of participants with a serious adverse event, regardless of causality, by dose and treatment
Number of Participants with One or More Serious Adverse Events (Part B) | Baseline up to approximately 50 days
  Number of participants with a serious adverse event, regardless of causality, by dose and treatment
Number of Participants with One or More Serious Adverse Events (Part C) | Baseline up to approximately 73 days
  Number of participants with a serious adverse event, regardless of causality, by dose and treatment

SECONDARY OUTCOMES:
Change from Baseline in Triplicate 12-lead Electrocardiogram (ECG) in Part A | Baseline up to 24 hours post-dose on day 2
  Mean change from baseline in triplicate 12-lead electrocardiogram (ECG)
Change in Baseline in Triplicate 12-lead ECG in Part B | Baseline up to 24 hours post-dose on day 6
  Mean change from baseline in triplicate 12-lead ECG
Change in Baseline in Triplicate 12-lead ECG in Part C | Baseline up to approximately day 28
  Mean change from baseline in triplicate 12-lead ECG
Change from Baseline in Single 12-Lead ECG in Part A | Baseline up to approximately 45 days
  Mean change from baseline in single 12-lead ECG
Change from Baseline in Single 12-Lead ECG in Part B | Baseline up to approximately 50 days
  Mean change from baseline in single 12-lead ECG
Change from Baseline in Single 12-Lead ECG in Part C | Baseline up to approximately 73 days
  Mean change from baseline in single 12-lead ECG
Number of Participants With Clinically Significant Changes in Vital Signs in Part A | Baseline up to approximately 45 days
  Respiration Rate, Heart Rate, Blood Pressure, Temperature
Number of Participants With Clinically Significant Changes in Vital Signs in Part B | Baseline up to approximately 50 days
  Respiration Rate, Heart Rate, Blood Pressure, Temperature
Number of Participants With Clinically Significant Changes in Vital Signs in Part C | Baseline up to approximately 73 days
  Respiration Rate, Heart Rate, Blood Pressure, Temperature
Number of participants with Physical Examination Findings in Part A | Baseline up to approximately 45 days
  Abnormal physical exam findings
Number of participants with Physical Examination Findings in Part B | Baseline up to approximately 50 days
  Abnormal physical exam findings
Number of participants with Physical Examination Findings in Part C | Baseline up to approximately 73 days
  Abnormal physical exam findings
Number of participants with Laboratory Test Results outside of reference range in Part A | Baseline up to approximately 45 days
  Laboratory results outside of reference range
Number of participants with Laboratory Test Results outside of reference range in Part B | Baseline up to approximately 50 days
  Laboratory results outside of reference range
Number of participants with Laboratory Test Results outside of reference range in Part C | Baseline up to approximately 73 days
  Laboratory results outside of reference range
Maximum Observed Drug Concentration (Cmax) in Part A | Baseline up to approximately 29 days
  Maximum observed plasma concentration of PRCL-02
Maximum Observed Drug Concentration (Cmax) in Part B | Baseline up to approximately 33 days
  Maximum observed plasma concentration of PRCL-02
Maximum Observed Drug Concentration (Cmax) in Part C | Baseline up to approximately 31 days
  Maximum observed plasma concentration of PRCL-02
Time to Maximum Drug Concentration (Tmax) in Part A | Baseline up to approximately 29 days
  Time to maximum plasma concentration of PRCL-02
Time to Maximum Drug Concentration (Tmax) in Part B | Baseline up to approximately 33 days
  Time to maximum plasma concentration of PRCL-02
Time to Maximum Drug Concentration (Tmax) in Part C | Baseline up to approximately 31 days
  Time to maximum plasma concentration of PRCL-02
Area Under the Plasma Concentration-Time Curve from Time 0 to Infinity (AUC0-∞) in Part A | Baseline up to approximately 29 days
  Area under the plasma concentration-time curve from time 0 to infinity
Area Under the Plasma Concentration-Time Curve During the Dosing Interval (24h) (AUC0-tau) in Part B | Baseline up to approximately 33 days
  Area under the plasma concentration-time curve during the dosing interval of 24 hours (24h)
Area Under The Plasma Concentration-Time Curve During the Dosing Interval (24h) (AUC0-tau) in Part C | Baseline up to approximately 31 days
  Area under the plasma concentration-time curve during the dosing interval (24h)
Minimum or Trough Concentration (Cmin) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Minimum or trough concentration of PRCL-02
Lag Time: Time Delay Between Drug Administration and First Observed Plasma Concentration (Tlag) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Time delay between administration of PRCL-02 and first observed plasma concentration
Elimination Rate (Ke) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Elimination rate of PRCL-02
Terminal Elimination Half-Life (t1/2) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Terminal elimination half-life of PRCL-02
Area Under the Plasma Concentration Time Curve from Time Zero to 24 Hours Post-dose (AUC0-24) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Area under the plasma concentration time curve from time zero to 24 hours
Area Under the Plasma Concentration Time Curve from Time Zero to the Last Observed Time Point (AUC0-t) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Area under the plasma concentration time curve from time zero to the last observed time point
Apparent Clearance (CL/F) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Apparent clearance of PRCL-02
Apparent Volume of Distribution (Vd/F) | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Apparent volume of distribution of PRCL-02
Accumulation Ratio | Predose up to approximately 29 days (Part A); 33 days (Part B), 31 days (Part C)
  Accumulation ratio of PRCL-02

CONTACTS AND LOCATIONS:
Overall Officials: Email PRCL@Choruspharma.com, Study Director — PRCL Research Inc.
Locations (6):
- Canada (6):
  - Dr. Chih-ho Hong Medical Inc, Surrey, British Columbia
  - Lynde Centre for Dermatology, Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - K Papp Clinical Research, Waterloo, Ontario
  - Centre de Dermatologie et Chirurgie Dermatologique, Montreal, Quebec
  - InVentiv Health, Québec

IPD SHARING:
Plan to Share IPD: No